CLINICAL TRIAL: NCT05710445
Title: Augmented Reality Heads-up Display to Improve Ultrasound Guided IV Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll subjects.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ali Dhanaliwala, Physician, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 852551
Record Dates: First submitted 2023-01-09; First posted 2023-02-02 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Phlebotomy
Keywords: Catheters; Augmented Reality; Ultrasound

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two groups. In the first group intravenous catheters will be placed per standard of care. In the second group, the catheter will be placed while the physicians utilizes augmented reality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality (Experimental): Subjects in this group will have their intravenous catheter placed while the physician uses a mixed reality headset to view the ultrasound images being used to guide the catheter placement.
  Interventions: Other: Augmented Reality
- Control (No Intervention): Subjects in this group will have their intravenous catheter placed using standard of care. The physician will use the monitor on the ultrasound machine only to view the ultrasound images being used to guide the catheter placement.

INTERVENTIONS:
Other: Augmented Reality — Mixed reality smart glasses will be used to view a virtual monitor which mirrors the ultrasound screen in real-time.
  Other Names: Microsoft HoloLens
  Arms: Augmented Reality

SUMMARY:
The purpose of this study is to assess the utility of an augmented reality headset for visualization of ultrasound images during ultrasound guided placement of an intravenous catheter.

DETAILED DESCRIPTION:
After being informed about the study, patients who require image guided intravenous access and give consent will have their intravenous catheter placed by a physician wearing mixed reality smart glasses. The mixed reality smart glasses will have an application that allows the physician to view the ultrasound images in a virtual monitor. The physician will then use the images viewed on this virtual monitor to guide placement of the intravenous catheter.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Referral for US assisted placement

Exclusion Criteria:

- Urgent/emergent requirement for IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Cannulation rate | At end of procedure, on average 30 minutes
  Number of successful venous cannulations as evaluated by treating physician

SECONDARY OUTCOMES:
Cannulation attempts | At end of procedure, on average 30 minutes
  Number of attempts needed to achieve a successful procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ali H Dhanaliwala, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.